CLINICAL TRIAL: NCT04412109
Title: Effect of Normal Saline Injection Volume on Epidural Pressure and Optic Nerve Sheath Diameter
Brief Title: Optic Nerve Sheath Diameter Difference Between Different Injection Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-01-081
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Optic Nerve Sheath Diameter
Keywords: Optic Nerve Sheath Diameter, Different volume

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- injection of low volume of saline (Active Comparator): low volume (5 cc) saline injection during thoracic epidural catheterization
  Interventions: Procedure: thoracic epidural catheterization
- injection of intermediate volume of saline (Active Comparator): intermediate volume (10 cc) saline injection during thoracic epidural catheterization
  Interventions: Procedure: thoracic epidural catheterization
- injection of high volume of saline (Active Comparator): high volume (20 cc) saline injection during thoracic epidural catheterization
  Interventions: Procedure: thoracic epidural catheterization

INTERVENTIONS:
Procedure: thoracic epidural catheterization — thoracic epidural catheterization for postoperative pain control

SUMMARY:
Valid method of indirect measurement of intracranial pressure is using optic nerve sheath diameter. Different volume of injection is known to affect the degree of increase of intracranial pressure.

This study is desinged to measure the changes of optic nerve sheath diameter and cerebral oxygenation when different volume of normal saline was injected.

DETAILED DESCRIPTION:
Previous study showed that different volume of injections (1.0 ml/kg vs. 1.5 ml/kg) during caudal anesthesia showed siginifiant increase of optic nerve sheath diameter in group of high volumes. Increase of ICP can result in harmful effect including reduced cerebral flow and oxygen saturation. Also, increase of ICP can cause headache, syncope and transient loss of visual acuity. The proven and valid method of measuring ICP indirectly is using optic nerve sheath diameter.

This study was designed to examine the changes of optic nerve sheath diameter and cerebral oxygenation when different volume of normal saline was injected.

ELIGIBILITY:
Inclusion Criteria:

* lung cancer
* liver cancer
* stomach cancer
* pancreas cancer
* gallbladder cancer

Exclusion Criteria:

* coagulopathy
* infection
* previous spine fusion at thoracic level
* previous brain lesion causing increased intracranial pressure

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
optic nerve sheath change during 4 time period | Baseline, 10 minutes, 20 minutes, 40 minutes after the completion of the intervention
  optic nerve sheath change during 4 time period using ultrasound

SECONDARY OUTCOMES:
cerebral oxygenation change during 4 time period | Baseline, 10 minutes, 20 minutes, 40 minutes after the completion of the intervention
  cerebral oxygenation change during 4 time period using pressure monitoring kit

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hee Hong, PhD, Principal Investigator — Keimyung University
Locations (1):
- Hong ji HEE, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong J, Kim JS, Lee YH. The Effect of Normal Saline Injection Volumes on the Optic Nerve Sheath Diameter during Thoracic Epidural Analgesia. Pain Physician. 2021 Nov;24(7):E1007-E1013. PMID 34704711